CLINICAL TRIAL: NCT02356575
Title: Choosing Options for Insomnia in Cancer Effectively (CHOICE): A Comparative Effectiveness Trial of Acupuncture and Cognitive Behavior Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-947
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Insomnia; Cancer
Keywords: surgery; chemotherapy; radiation; Acupuncture; 16-947
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms | interventions — Acupuncture Therapy; Cognitive Behavioral Therapy

ARMS (2):
- Acupuncture Group (Active Comparator): In the acupuncture group, patients will receive ten treatments of acupuncture over eight weeks.
  Interventions: Other: Acupuncture
- CBT-I Group (Active Comparator): In the CBT-I group, patients will receive seven sessions of CBT-I over eight weeks.
  Interventions: Other: Cognitive Behavior Therapy

INTERVENTIONS:
Other: Acupuncture
  Arms: Acupuncture Group
Other: Cognitive Behavior Therapy
  Arms: CBT-I Group

SUMMARY:
The aim of this study is to determine which of two treatments (acupuncture or cognitive behavioral therapy) works better for treating insomnia in cancer survivors. The investigator also wants to study the factors that might impact why someone might prefer or do better in one treatment over the other.

Group 1 will get Acupuncture - Acupuncture is an ancient Chinese Technique of using very thin needles inserted in the skin to treat different symptoms and illness, and to promote healing.

Group 2 will get Cognitive Behavioral Therapy for Insomnia (CBT-I) - CBT-I is a treatment to address behaviors and thoughts that are known to effect problems with sleep.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking, age ≥ 18 years old
* A diagnosis of cancer with no restrictions placed on type of cancer or stage. Eligibility criteria are not be restricted to MSK confirmed biopsy/diagnosis. Participating institution's testing is sufficient for other study sites.
* Completed active treatment (surgery, chemotherapy, and/or radiotherapy) at least one month prior to study initiation (patients on continued hormone treatment or maintenance targeted therapies will not be excluded).
* A score >7 on our primary outcome (the Insomnia Severity Index)
* A diagnosis of insomnia disorder as defined by the Diagnostic and Statistical Manual of Mental disorders, 5th Edition (DSM-5), per the diagnostic interview. According to this nosology, insomnia is defined as dissatisfaction with sleep quality or quantity characterized by difficulty initiating sleep, maintaining sleep, or early morning awakenings that cause significant distress or impairment in daytime functioning and occur at least three nights per week for at least three months despite adequate opportunity for sleep.
* Patients using psychotropic medication (e.g. antidepressants) will remain eligible for study participation provided that the dose was not recently altered (stable over the previous 6-weeks).
* Patients using hypnotics or sedatives will be eligible for study participation. Considering the high use of benzodiazepines within the oncology population, past research has included participants who met diagnostic criteria for insomnia, despite the use of benzodiazepines, and included monitoring of medication use.

Exclusion Criteria:

* Another sleep disorder, other than sleep apnea, that is not adequately treated.
* Previous experience with CBT or acupuncture to treat insomnia
* Currently participating in another acupuncture trial or a trial to treat insomnia
* The presence of another Axis I disorder not in remission
* Employment in a job requiring shift work that would impair the ability to establish a regular sleep schedule
* Patients who are currently taking oral (not including oral sprays/inhalers) or intravenous corticosteroids as part of treatment for cancer or any other condition will be excluded because of the potential of these drugs to induce insomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Li Y, Liou KT, Schofield E, Atkinson TM, Mao JJ. Novel bayesian nonparametric unsupervised learning approach to precision symptom management in cancer survivors: a re-analysis of a comparative effectiveness trial. J Behav Med. 2026 Jan 23. doi: 10.1007/s10865-025-00621-7. Online ahead of print. PMID 41575714
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Kwag E, Li X, Garland S, Bryl K, Taylor L, Li QS, Amann L, Mao JJ, McConnell KM. Acupuncture versus cognitive behavioral therapy for anxiety among cancer survivors with insomnia: An exploratory analysis of a randomized clinical trial. Integr Med Res. 2025 Dec;14(4):101213. doi: 10.1016/j.imr.2025.101213. Epub 2025 Aug 7. PMID 40896348
- [Derived] Liou KT, Garland SN, Li QS, Sadeghi K, Green J, Autuori I, Orlow I, Mao JJ. Effects of acupuncture versus cognitive behavioral therapy on brain-derived neurotrophic factor in cancer survivors with insomnia: an exploratory analysis. Acupunct Med. 2021 Dec;39(6):637-645. doi: 10.1177/0964528421999395. Epub 2021 Mar 22. PMID 33752446
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture Group: In the acupuncture group, patients will receive ten treatments of acupuncture over eight weeks.
  Acupuncture
- CBT-I Group: In the CBT-I group, patients will receive seven sessions of CBT-I over eight weeks.
  Cognitive Behavior Therapy
Period: Overall Study
Arm/Group | Acupuncture Group | CBT-I Group
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture Group | CBT-I Group | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Full Range); unit: years] | 62.3 [27.5 to 86.3] | 60.7 [31 to 79.8] | 61.5 [27.5 to 86.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 37 | 32 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 77 | 75 | 152
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 27 | 44
  White | 61 | 52 | 113
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI) at Baseline
Description: The Insomnia Severity Index (ISI) is one of the few well-validated patient-reported outcome measure designed to specifically assess the impact on daytime functioning and the amount of associated distress. The ISI includes 7 items that are scored on a five-point scale ranging from 0 to 4 with higher scores representing more severe insomnia symptoms. The optimal cutoff scores are 0-7 (no clinically significant sleep difficulties), 8-14 (sleep difficulties warrant further investigation), and 15+ (presence of clinically significant insomnia). Maximum score on this scale is 28.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
score on a scale | 17.6 (4.1) | 18.5 (4.4)

2. Primary Outcome: Insomnia Severity Index (ISI) Change From Baseline at 8 Weeks
Description: A greater negative value represents improvement in symptoms.
  The Insomnia Severity Index (ISI) is one of the few well-validated patient-reported outcome measure designed to specifically assess the impact on daytime functioning and the amount of associated distress. The ISI includes 7 items that are scored on a five-point scale ranging from 0 to 4 with higher scores representing more severe insomnia symptoms. The optimal cutoff scores are 0-7 (no clinically significant sleep difficulties), 8-14 (sleep difficulties warrant further investigation), and 15+ (presence of clinically significant insomnia). Maximum score on this scale is 28.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -8.31 [-9.36 to -7.26] | -10.91 [-11.97 to -9.85]

3. Primary Outcome: Insomnia Severity Index (ISI) Change From Baseline at 20 Weeks
Description: as for outcome 2
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -8.59 [-9.65 to -7.55] | -11.12 [-12.19 to -10.06]

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) at Baseline
Description: The Pittsburgh Sleep Quality Index was specifically designed for use in clinical populations to assess seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction) and a global score. It consists of 19 self-rated questions that are scored on a 0 to 3 scale over a period of one month, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of 5 or greater indicates a "poor" sleeper. Overall score ranges from 0 to 21.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 11.8 (3.2) | 12.1 (3.7)

5. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Change From Baseline at 8 Weeks
Description: A greater negative value represents improvement in symptoms. Please note this is the change in score from baseline at 8 weeks.
  The Pittsburgh Sleep Quality Index was specifically designed for use in clinical populations to assess seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction) and a global score. It consists of 19 self-rated questions that are scored on a 0 to 3 scale over a period of one month, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of 5 or greater indicates a "poor" sleeper. Overall score ranges from 0 to 21.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -4.39 [-5.10 to -3.67] | -5.90 [-6.61 to -5.18]

6. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) From Baseline at 20 Weeks
Description: A greater negative value represents improvement in symptoms. Please note that this is the change in score from baseline to 20 weeks.
  The Pittsburgh Sleep Quality Index was specifically designed for use in clinical populations to assess seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction) and a global score. It consists of 19 self-rated questions that are scored on a 0 to 3 scale over a period of one month, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of 5 or greater indicates a "poor" sleeper. Overall score ranges from 0 to 21.
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -4.62 [-5.33 to -3.91] | -5.84 [-6.56 to -5.13]

7. Secondary Outcome: The Consensus Sleep Diary (CSD) Baseline Sleep Onset
Description: The Consensus Sleep Diary (CSD) will be used to calculate sleep onset at baseline. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | 32.1 (29.3) | 47.1 (62.1)

8. Secondary Outcome: The Consensus Sleep Diary (CSD) Sleep Onset Change From Baseline at Week 8
Description: A greater negative value represents improvement in symptoms. Please note this is the change in sleep onset from Baseline at Week 8.
  The Consensus Sleep Diary (CSD) will be used to calculate sleep onset. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | -10.80 [-16.46 to -5.14] | -27.13 [-33.12 to -21.14]

9. Secondary Outcome: The Consensus Sleep Diary (CSD) Sleep Onset Change From Baseline at Week 20
Description: A greater negative value represents improvement in symptoms. Please note this is the change in sleep onset from Baseline at Week 20.
  The Consensus Sleep Diary (CSD) will be used to calculate sleep onset. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | -10.91 [-16.70 to -5.13] | -24.37 [-30.36 to -18.38]

10. Secondary Outcome: The Consensus Sleep Diary (CSD) Minutes Wake After Sleep Onset at Baseline
Description: The Consensus Sleep Diary (CSD) will be used to calculate wake after sleep onset. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | 58.0 (38.8) | 53.6 (42.1)

11. Secondary Outcome: The Consensus Sleep Diary (CSD) Minutes Wake After Sleep Onset Change From Baseline at Week 8
Description: A greater negative value represents improvement in symptoms. Please note this is the change from Baseline to Week 8.
  The Consensus Sleep Diary (CSD) will be used to calculate sleep-onset latency. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | -26.89 [-34.16 to -19.61] | -35.83 [-43.51 to -28.16]

12. Secondary Outcome: The Consensus Sleep Diary (CSD) Minutes Wake After Sleep Onset Change From Baseline at 20 Weeks
Description: A greater negative value represents improvement in symptoms. Please note this is the change from Baseline to Week 20.
  The Consensus Sleep Diary (CSD) will be used to calculate sleep-onset latency. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | -22.01 [-29.45 to -14.58] | -29.51 [-37.16 to -21.87]

13. Secondary Outcome: The Consensus Sleep Diary (CSD) Baseline Total Sleep Time
Description: The Consensus Sleep Diary (CSD) will be used to calculate total sleep time. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | 346.1 (82.1) | 340.8 (99.2)

14. Secondary Outcome: The Consensus Sleep Diary (CSD) Total Sleep Time Change From Baseline at Week 8
Description: A greater positive value represents improvement in symptoms. Please note this reflects the change from Baseline to Week 8.
  The Consensus Sleep Diary (CSD) will be used to calculate total sleep time. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | 61.81 [45.79 to 77.84] | 35.01 [18.12 to 51.91]

15. Secondary Outcome: The Consensus Sleep Diary (CSD) Total Sleep Time Change From Baseline at Week 20
Description: A greater positive value represents improvement in symptoms. Please note this reflects the change from Baseline to Week 20.
  The Consensus Sleep Diary (CSD) will be used to calculate total sleep time. Sleep diaries are considered a reliable and valid patient report of nightly insomnia symptoms. Participants will complete the sleep diary daily throughout treatment.
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
minutes | 50.71 [34.39 to 67.03] | 45.23 [28.33 to 62.12]

16. Secondary Outcome: The Consensus Sleep Diary (CSD) Sleep Efficiency at Baseline
Description: Sleep efficiency was calculated as a ratio of total sleep time divided by time in bed multiplied by 100 to yield a percentage. A higher number indicates better sleep efficiency.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of efficiency
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
percentage of efficiency | 73.2 (13.5) | 72.1 (18.3)

17. Secondary Outcome: The Consensus Sleep Diary (CSD) Sleep Efficiency Change From Baseline at Week 8
Description: A greater positive value represents improvement in symptoms. Please note this reflects a change from Baseline to Week 8.
  Sleep efficiency was calculated as a ratio of total sleep time divided by time in bed multiplied by 100 to yield a percentage. higher number indicated better sleep efficiency.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
percentage change | 0.11 [0.08 to 0.13] | 0.16 [0.13 to 0.18]

18. Secondary Outcome: The Consensus Sleep Diary (CSD) Sleep Efficiency Change From Baseline at Week 20
Description: A greater positive value represents improvement in symptoms. Please note this reflects a change from Baseline to Week 20.
  Sleep efficiency was calculated as a ratio of total sleep time divided by time in bed multiplied by 100 to yield a percentage. higher number indicated better sleep efficiency.
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
percentage change | 0.10 [0.07 to 0.12] | 0.13 [0.10 to 0.16]

19. Secondary Outcome: Brief Pain Inventory (BPI) at Baseline
Description: Brief Pain Inventory (BPI) is an 11-item pain assessment tool for use with cancer patients. The BPI has two subscales, pain severity and pain interference. Here we reported BPI severity which is an average of 4 questions. The BPI severity score ranges from 0-10 with higher number indicating worse pain symptom.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 2.4 (2.4) | 2.1 (2.0)

20. Secondary Outcome: Brief Pain Inventory (BPI) Change From Baseline at Week 8
Description: A greater negative value represents improvement in symptoms.
  Brief Pain Inventory (BPI) is an 11-item pain assessment tool for use with cancer patients. The BPI has two subscales, pain severity and pain interference. Here we reported BPI severity which is an average of 4 questions. The BPI severity score ranges from 0-10 with higher number indicating worse pain symptom.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -0.49 [-0.81 to -0.16] | 0.00 [-0.33 to 0.33]

21. Secondary Outcome: The Brief Pain Inventory (BPI) Change From Baseline at Week 20
Description: as for outcome 20
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -0.46 [-0.79 to -0.14] | -0.35 [-0.68 to -0.02]

22. Secondary Outcome: Multidimensional Fatigue Inventory-Short Form (MFSI-SF) at Baseline
Description: The Multidimensional Fatigue Inventory-Short Form (MFSI-SF) is a 30 item self-report measure. Higher scores indicate more fatigue.
  A 30 item self-report measure comprised of five subscales (general, emotional, physical, mental, vigor) and a total fatigue score. We reported the total fatigue score by summing all the items. Multidimensional Fatigue Inventory-Short Form / MFSI-SF total score ranges from 0 to 120 with higher score indicates more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 19.8 (21.3) | 21.9 (22.3)

23. Secondary Outcome: Multidimensional Fatigue Inventory-Short Form (MFSI-SF) Change From Baseline at Week 8
Description: A greater negative value represents improvement in symptoms.
  A 30 item self-report measure comprised of five subscales (general, emotional, physical, mental, vigor) and a total fatigue score. We reported the total fatigue score by summing all the items. Multidimensional Fatigue Inventory-Short Form / MFSI-SF total score ranges from 0 to 120 with higher score indicates more fatigue.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -10.82 [-13.94 to -7.70] | -12.48 [-15.69 to -9.27]

24. Secondary Outcome: Multidimensional Fatigue Inventory-Short Form (MFSI-SF) Change From Baseline at Week 20
Description: as for outcome 23
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: score on MFSI-F
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
score on MFSI-F | -12.20 [-15.32 to -9.08] | -11.19 [-14.38 to -8.00]

25. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety at Baseline
Description: This is a 14 item, self-rated instrument for anxiety (7 items) and depression (7 items) symptoms in the past week and has been extensively used in people with cancer. Established cutoffs for the depression and anxiety scales are independent and are: 0-7 not significant; 8-10 subclinicao; and 11-21 clinically significant depression/anxiety.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 7.8 (4.0) | 7.8 (4.3)

26. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Change in Anxiety From Baseline at Week 8
Description: A greater negative value represents improvement in symptoms.
  This is a 14 item, self-rated instrument for anxiety (7 items) and depression (7 items) symptoms in the past week and has been extensively used in people with cancer. Established cutoffs for the depression and anxiety scales are independent and are: 0-7 not significant; 8-10 subclinical; and 11-21 clinically significant depression/anxiety.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -2.21 [-2.82 to -1.60] | -1.93 [-2.56 to -1.30]

27. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Change in Anxiety From Baseline at Week 20
Description: as for outcome 26
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -1.94 [-2.55 to -1.33] | -1.83 [-2.46 to -1.20]

28. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Depression at Baseline
Description: This is a 14 item, self-rated instrument for anxiety (7 items) and depression (7 items) symptoms in the past week and has been extensively used in people with cancer. Established cutoffs for the depression and anxiety scales are independent and are: 0-7 not significant; 8-10 subclinical; and 11-21 clinically significant depression/anxiety.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 4.6 (3.1) | 5.1 (3.4)

29. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Change in Depression From Baseline at Week 8
Description: as for outcome 26
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -1.06 [-1.57 to -0.55] | -1.45 [-1.98 to -0.92]

30. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Change in Depression From Baseline at Week 20
Description: as for outcome 26
Time Frame: 20 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | -0.91 [-1.42 to -0.40] | -1.22 [-1.75 to -0.69]

31. Secondary Outcome: Global Physical Health Scale (PROMIS® Global 10) at Baseline
Description: The 10-item Patient-Reported Outcomes Measurement Information System Global Health Scale (PROMIS® Global 10) was used to assess key quality of life domains including pain, fatigue, mental health, physical health, social health, and overall health. There are two 4-item domains: global physical health (domain score ranges from 4 to 20) and global mental health (domain score ranges from 4 to 20). Higher score indicates better quality of life. A greater positive value represents improvement in symptoms from baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 45.2 (8.4) | 43.4 (8.7)

32. Secondary Outcome: Global Physical Health Scale (PROMIS® Global 10) Change From Baseline at Week 8
Description: A greater positive value represents improvement in symptoms.
  The 10-item Patient-Reported Outcomes Measurement Information System Global Health Scale (PROMIS® Global 10) was used to assess key quality of life domains including pain, fatigue, mental health, physical health, social health, and overall health. There are two 4-item domains: global physical health (domain score ranges from 4 to 20) and global mental health (domain score ranges from 4 to 20). Higher score indicates better quality of life. A greater positive value represents improvement in symptoms from baseline.
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 2.19 [0.92 to 3.46] | 3.73 [2.44 to 5.02]

33. Secondary Outcome: Global Physical Health Scale (PROMIS® Global 10) Change From Baseline at Week 20
Description: as for outcome 32
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 3.29 [2.02 to 4.56] | 4.49 [3.20 to 5.78]

34. Secondary Outcome: Global Mental Health Scale (PROMIS® Global 10) at Baseline
Description: as for outcome 31
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 45.0 (8.0) | 44.1 (8.2)

35. Secondary Outcome: Global Mental Health Scale (PROMIS® Global 10) Change From Baseline at Week 8
Description: as for outcome 32
Time Frame: 8 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 3.34 [1.99 to 4.69] | 3.39 [2.02 to 4.76]

36. Secondary Outcome: Global Mental Health Scale (PROMIS® Global 10) Change From Baseline at Week 20
Description: as for outcome 32
Time Frame: 20 weeks from baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 4.08 [2.73 to 5.43] | 3.29 [2.04 to 4.78]

37. Secondary Outcome: Treatment Expectancy Scale: Expectancy for CBT-I Treatment
Description: A 4-item instrument that measures treatment expectancy. The total score was calculated by summing all 4 items. Score ranges from 4 to 20 with higher score indicates greater treatment expectancy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 12.8 (3.5) | 13.2 (2.9)

38. Secondary Outcome: Treatment Expectancy Scale: Expectancy for Acupuncture Treatment
Description: as for outcome 37
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture Group | CBT-I Group
Number analyzed (Participants) | 80 | 80
units on a scale | 13.3 (4.0) | 13.2 (3.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Acupuncture Group | CBT-I Group
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 10/80 | 5/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture Group (N=80) | CBT-I Group (N=80)
Soreness at needling site (General disorders) | 5 | 0
Dizziness (Nervous system disorders) | 2 | 0
Drowsiness (Nervous system disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Bruising at needling site (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Itchiness at needling site (General disorders) | 1 | 0
Pain at needling site (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT02356575/Prot_SAP_000.pdf